CLINICAL TRIAL: NCT06092645
Title: An Open-label, Single-arm, Multicenter, Phase II Clinical Study of Surufatinib Plus Cadonilimab as Second-line Therapy in Patients With Unresectable or Metastatic Bile Duct Adenocarcinoma
Brief Title: Surufatinib Plus Cadonilimab in Patients With Unresectable or Metastatic Bile Duct Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ying Jieer, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2023-386
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Bile Duct Adenocarcinoma
MeSH Terms: interventions — surufatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- surufatinib plus Cadonilimab (Experimental): Surufatinib: 250mg , po,qd, d1-d21, every 3 weeks for a treatment cycle. Cardonilimab: 10mg/kg, iv, d1, every 3 weeks for a treatment cycle
  Interventions: Drug: surufatinib plus cadonilimab

INTERVENTIONS:
Drug: surufatinib plus cadonilimab — Surufatinib: 250mg , po,qd, d1-d21, every 3 weeks for a treatment cycle. Cadonilimab: 10mg/kg, iv, d1, every 3 weeks for a treatment cycle
  Other Names: surufatinib plus AK104

SUMMARY:
This is an open-label, single-arm, multicenter Phase II clinical study to evaluate the efficacy and safety of surufatinib combined with cardanilimab in second-line treatment of patients with inoperable or metastatic bile duct adenocarcinoma

DETAILED DESCRIPTION:
This is an open-label, single-arm, multicenter Phase II clinical trial. It is planned to enroll patients with inoperable or metastatic bile duct adenocarcinoma who have progressed through first-line chemotherapy combined with immunotherapy in several hospitals across the country to evaluate the efficacy and safety of second-line treatment with surufatinib Combination With Cadonilimab.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate in the study and sign the informed consent;
2. Over 18 years old (including 18 years old), regardless of gender;
3. Expected survival ≥12 weeks;
4. Within 7 days before the first administration of the study drug, the ECOG physical status score was 0 or 1;
5. Locally advanced or metastatic cholangiocarcinoma (including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder carcinoma) that is histologically and/or cytologically confirmed and is incurable and unresectable;
6. The investigator confirmed the presence of at least one measurable lesion according to RECIST 1.1 criteria. Target lesions located within the field of prior radiotherapy or within the area following local treatment are considered measurable if they demonstrate progression.
7. Patients who have Progression after first-line chemotherapy combined with PD-1/L1 inhibitors for advanced unresectable or metastatic bile duct adenocarcinoma
8. Adequate organ function 1) Blood routine examination: (no transfusion within 14 days prior to screening, no use of granulocyte colony stimulating factor [G-CSF], no use of drug correction) : i. Neutrophils ≥1.5×109/L; ii. Platelet ≥75×109/L; iii. Hemoglobin ≥90g/L; 2) Biochemical examination: (no albumin infusion within 14 days prior to screening) : iv. Serum creatinine ≤1.5× upper limit of normal (ULN), or creatinine clearance > 50 mL/min; v. Serum total bilirubin ≤1.5×ULN (subjects with Gilbert syndrome allow total bilirubin ≤3×ULN); vi. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2.5×ULN; In subjects with liver metastasis, ALT and AST≤5×ULN; 3) Coagulation function: vii. International Standardized Ratio (INR) ≤2.3 or prothrombin time; (PT) exceeding the normal control range ≤6 seconds; 4) Urinary protein viii. Urinary protein < 2+ (If urine protein ≥2+, it can be performed for 24 hours (h) Urinary protein quantification, 24h urinary protein quantification < 1.0g can be included) 5) Heart function: ix. New York College of Cardiology (NYHA) rating < 3; x. Left ventricular ejection fraction ≥50%;
9. If the patient has active hepatitis B virus (HBV) infection: HBV-deoxyribonucleic acid (DNA) must be < 500 IU/mL (< 2500 copy/ml if the study center only has copy/ml testing units) and is willing to receive antiviral therapy throughout the study period; Hepatitis C virus (HCV) ribonucleic acid (RNA) positive patients must receive antiviral therapy according to standard local treatment guidelines and have liver function within CTCAE level 1 elevation;
10. The patient must have an appropriate nutritional status, i.e. body mass index(BMI) ≥ 18 kg/m2, body weight ≥ 40 kg, and serum albumin ≥ 3.0 g/dL.
11. Within 28 days prior to enrollment, women of reproductive age must confirm a negative serum pregnancy test and consent to effective contraceptive use during the study drug use period and within 60 days after the last dose. In this protocol, women of reproductive age are defined as sexually mature women: 1) who have not undergone hysterectomy or bilateral oophorectomy, 2) who have not had natural menstrual cessation for 24 consecutive months (amenorrhea after cancer treatment does not exclude fertility) (i.e., who have menstruated at any time during the previous 24 consecutive months); Female spouses of male subjects of childbearing age should also follow the above contraceptive requirements.

Exclusion Criteria:

Patients who meet any of the following conditions will not be admitted to the study:

1. Active malignancy other than bile duct malignancy within 5 years or at the same time. Localized tumors that have been cured, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder carcinoma, prostate carcinoma in situ, cervical carcinoma in situ, breast carcinoma in situ, etc.
2. Patients who are preparing for or have previously received an organ or allogeneic bone marrow transplant;
3. Moderate or severe ascites with clinical symptoms require therapeutic puncture or drainage (except those who only show a small amount of ascites without clinical symptoms on imaging); Uncontrolled or moderate or above pleural effusion and pericardial effusion;
4. Study a history of gastrointestinal bleeding or a definite tendency to gastrointestinal bleeding within 6 months before the start of treatment, such as: Patients with bleeding risk or severe esophageal and gastric varices, locally active digestive ulcer lesions, and persistent positive occult blood in stool could not be included in the group (if the stool was positive for occult blood at baseline, it could be re-examined; if the stool was still positive after re-examination, gastroduodenal microscopy (EGD) was required; if EGD suggested bleeding risk, esophageal and gastric varices could not be included in the group).
5. Known hereditary or acquired bleeding (e.g. coagulation disorders) or thrombotic tendencies, e.g. in hemophiliacs; Is currently or recently (within 10 days prior to the start of study therapy) used full dose oral or injectable anticoagulants or thrombolytic agents for therapeutic purposes (prophylactic use of low-dose aspirin, low-molecular weight heparin permitted);
6. Currently using or recently used (within 10 days before the start of study treatment) aspirin>325 mg/ day (maximum antiplatelet dose) or dipyridamole, ticlopidine, clopidogrel, and cilostazole;
7. Thrombosis or embolism events, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), pulmonary embolism, etc., occurred within 6 months before the start of the study treatment;
8. Have clinical symptoms or diseases of the heart that are not well controlled, such as:

1) According to the New York Heart Association (NYHA) standards for Grade II or higher cardiac insufficiency or cardiac color ultrasound: LVEF (left ventricular ejection fraction) <50%; 2) Unstable angina pectoris；3) Myocardial infarction occurred within 1 year before the start of study treatment；4) Clinically significant supraventricular or ventricular arrhythmias require treatment or intervention；5) QTc>450ms (male); QTc>470ms (female) (QTc interval calculated by Fridericia formula; If the QTc is abnormal, it can be detected three times at an interval of 2 minutes, and the average value is taken); 9. Have high blood pressure that is not well controlled by antihypertensive medication (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90 mmHg (based on the average of BP readings taken from ≥2 measurements), allowing the above parameters to be achieved with antihypertensive therapy; Hypertensive crisis or hypertensive encephalopathy in the past; 10. Major vascular disease (e.g., aortic aneurysms requiring surgical repair or recent peripheral arterial thrombosis) developed within 6 months prior to the start of study therapy; 11. Severe, unhealed or open wounds and active ulcers or untreated fractures; 12. Received major surgery within 4 weeks prior to the start of study treatment (except for diagnosis) or expected to require major surgery during the study period; 13. Inability to swallow tablets, malabsorption syndrome or any condition affecting gastrointestinal absorption； 14. Evidence of abdominal gas that cannot be explained by puncture or recent surgical procedures; 15. Past or current central nervous system metastasis; 16. Be suffering from uncontrolled systemic diseases, including diabetes mellitus, hypertension, pulmonary fibrosis, acute lung disease, interstitial lung disease, cirrhosis of the liver, angina pectoris, severe arrhythmia, etc.; 17. People with current or prior history of interstitial pneumonia or interstitial lung disease requiring hormone therapy, or other pulmonary fibrosis, institutional pneumonia (e.g., Subjects with bronchiolitis oblans), pneumoconiosis, drug-related pneumonia, idiopathic pneumonia, or with evidence of active pneumonia or severely impaired lung function on chest computed tomography (CT) images during screening were allowed to have radiation pneumonia in the radiation field; Active tuberculosis; 18. Presence of active autoimmune disease or history of autoimmune disease with possible recurrence (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, pituitaritis, vasculitis, nephritis, hyperthyroidism, hypothyroidism [subjects controllable by hormone replacement therapy only may be included]); Participants with non-systemic skin diseases such as vitiligo, psoriasis, and alopecia, controlled type 1 diabetes treated with insulin, or asthma in complete remission in childhood, were enrolled without any intervention as adults; Patients with asthma requiring medical intervention with bronchodilators were excluded; 19. Use of immunosuppressants or systemic hormone therapy for immunosuppressive purposes within 14 days prior to initiation of study therapy (dose>10mg/day prednisone or other equivalent hormone); 20. Use of strong CYP3A4/ CYP2C19 inducers including rifampicin (and its analogues) and hypericum perforatum or strong CYP3A4/ CYP2C19 inhibitors within 14 days prior to initiation of study therapy; 21. Known to have a history of severe allergy to any monoclonal antibody or anti-angiogenesis targeting drug; 22. Severe infections, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia, in the 4 weeks prior to initiation of study treatment; Oral or intravenous administration of therapeutic antibiotics within 2 weeks prior to starting study treatment (patients receiving prophylactic antibiotics (for example, to prevent urinary tract infections or exacerbations of COPD) are eligible for study participation； 23. Patients with congenital or acquired immune deficiency (such as HIV infection); 24. Prior treatment with other immunosuppressants (other than PD-1/L1 inhibitors) or prior treatment with tyrosine kinase inhibitors; 25. To permit palliative radiotherapy for non-target lesions to control symptoms, it must be completed at least 2 weeks prior to the initiation of study therapy, and radiation-related adverse events have not recovered to ≤CTCAE grade 1; 26. Has received live attenuated vaccines within 28 days prior to initiation of study treatment, or is expected to require such vaccines during treatment with cardonilizumab or within 60 days after the last administration of cardonilizumab; 27. Received anti-tumor cytotoxic drug therapy, biologic drug therapy (such as monoclonal antibodies), immunotherapy (such as interleukin-2 or interferon), or other investigational drug therapy within 4 weeks prior to study enrollment; 28. According to the investigator's judgment, the patient has other factors that may affect the study results or lead to the forced termination of the study, such as alcoholism, drug abuse, other serious diseases (including mental illness) requiring combined treatment, serious laboratory abnormalities, and family or social factors, which will affect the safety of the patient.

29. The toxicity of previous antitumor therapy has not returned to CTCAE level 0-1, except in the following cases:

1. hair loss;
2. Pigmentation;
3. Peripheral nerve toxicity has returned to <CTCAE Level 2;
4. Long-term toxicity caused by radiotherapy, which could not be recovered according to the investigators; 30. Subjects with active tuberculosis (TB) who are receiving anti-TB therapy or have received anti-TB therapy within 1 year prior to screening; 31. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 12 months
  Refers to the date from the date of admission to the date of the first progression of disease or death of any cause, using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).

SECONDARY OUTCOMES:
Overall survival (OS) | up to 36 months
  The time interval between the start date of study drug and the date of death (any cause)
Objective response rate(ORR) | up to 12 months
  The number of cases in which tumor size is reduced to PR or CR / the total number of evaluable cases (%)
Disease control rate (DCR) | up to 12 months
  Percentage of confirmed cases including complete remission (CR), partial remission (PR) and disease stability (SD) among patients with evaluable efficacy
Incidence of adverse events | Until the last medication for 30 days (±7 days) or before the start of other anti-tumor therapy (whichever occurs first)
  Categorized according to NCI Common Toxicity Criteria version 5.0. Summarized in terms of type, severity (grade 1-5), and dose level in tabular format.

CONTACTS AND LOCATIONS:
Overall Officials: Jieer Ying, M.D., Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China